CLINICAL TRIAL: NCT06329544
Title: The Effects of a High Fructose Diet on the Gut Microbiome and Metabolic Health: A Controlled Clinical Intervention Study
Brief Title: High Fructose Diet, the Gut Microbiome, and Metabolic Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Metabolic Solutions Inc. (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ryan Walker, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY-23-01572; 1R01DK137968-01 (NIH)
Record Dates: First submitted 2024-03-18; First posted 2024-03-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: MASLD; Type 2 Diabetes; Obesity
Keywords: Microbiome; MASLD; Obesity; Fructose; Fatty Liver
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Fatty Liver | interventions — Fructose; Glucose

STUDY DESIGN:
Intervention Model Description: The study will be a double-blinded (participants and select study personnel), randomized controlled crossover dietary intervention design.
Who Masked: Participant, Investigator
Masking Description: All participants undergo both treatment arms but will be blinded to the order.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fructose Dietary then Glucose Dietary (Experimental): Participants that will be randomized to the 12-day isocaloric weight-maintaining high fructose diet, then will change to the 12-day isocaloric weight-maintaining high glucose diet after a 10-day washout period.
  Interventions: Dietary Supplement: Fructose; Dietary Supplement: glucose
- Glucose Dietary then Fructose Dietary (Experimental): Participants that will be randomized to the 12-day isocaloric weight-maintaining high glucose diet, then will change to the12-day isocaloric weight-maintaining high fructose diet after a 10-day washout period.
  Interventions: Dietary Supplement: Fructose; Dietary Supplement: glucose

INTERVENTIONS:
Dietary Supplement: Fructose — 12-day isocaloric weight-maintaining high fructose diet (25% total calories from added fructose)
Dietary Supplement: glucose — 12-day isocaloric weight-maintaining high glucose diet (25% total calories from added glucose)

SUMMARY:
Americans commonly consume excess amounts of dietary fructose. Added fructose has been shown to have an adverse impact on metabolic health, including increased insulin resistance and type 2 diabetes (T2D) risk. However, the mechanisms that link dietary fructose and metabolic health are poorly understood. Malabsorption or incomplete metabolism of fructose in the small intestine is common in the population. Excess fructose reaches the colon where it may change the structure and function of the gut microbiome, alter bacterial metabolites and trigger inflammatory responses impacting T2D risk. To elucidate whether commonly consumed levels of dietary fructose influence metabolic outcomes through altering the gut microbiome, the research team will randomize 30 participants to a controlled cross-over dietary intervention, in which the participants will consume 12-day isocaloric, added fructose or glucose diets (25% of total calories) separated by a 10-day controlled diet washout period.

The research team aims to:

1. Determine the relationships between high fructose consumption, the gut microbiome and metabolic risk.
2. Characterize the causal role(s) that fructose-induced alterations to the gut microbiome have on metabolic risk using a germ-free mouse model.

The research team will measure 1) microbiota community structure and function via metagenomic sequencing of stool, 2) fecal metabolites via targeted and untargeted metabolomics, 3) anthropometrics, 4) insulin resistance, serum markers of T2D risk and inflammatory cytokines, 5) fecal microbial carbohydrate oxidation capacity and 6) liver fat via MRI elastography. The research team will use novel statistical approaches, including Distributed Lag Modeling, to understand the complex relationships between diet, the microbiome, metabolites and health outcomes.

The research team will then conduct controlled dietary interventions and fecal microbiome transplantation studies in germ-free mice. Donor fecal samples from human participants in both the glucose and fructose arms of the clinical intervention will be transplanted into germ-free and colonized mice to establish a causal relationship between fructose-induced changes to the gut microbiome, liver fat and metabolic and inflammatory changes known to increase risk for T2D.

The research team aims to comprehensively assess the structural and functional changes to the gut microbiome brought about by a high fructose diet. Determining the impact of excess fructose on the microbiome will help identify novel means by which fructose contributes to metabolic disease risk. In addition to identifying strategies to improve metabolic health in adults, data from this proposal could help inform targeted approaches to mitigate future disease risk in vulnerable populations that consume high levels of fructose, such as children.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be determined to be a fructose malabsorber (screening visit) via hydrogen breath test.

Exclusion Criteria:

* Use of probiotic/prebiotic/synbiotic supplements
* Consumption of > 1 sugar sweetened beverage per day
* Antibiotics within 3 months prior to enrollment or during intervention
* Vegetarian, vegan or other restrictive dietary habits
* Food allergy
* Alcohol consumption in excess of 2 drink per day

The following additional factors will be exclusion criteria:

* Physician diagnosis of a major medical illness (including type 1 or type 2 diabetes) or eating disorder
* Physical, mental, or cognitive handicaps that prevent participation
* Chronic use of any medication that may affect body weight or composition, insulin resistance, or lipid profiles;
* Current smoking (more than 1 cigarette in the past week) or use of other recreational drugs; e) restrictive dietary habits;
* food allergy;
* excess alcohol consumption;
* recent use of pro-, pre- or Synbiotics of receipt of antibiotics within 3 months prior to enrollment or during the intervention;
* consumption of greater than 1 sugar sweetened beverage per day prior to enrollment

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Liver proton density fat fraction (PDFF) | year 3
  Liver proton density fat fraction (PDFF) in %
Degree of fibrosis | year 3
  Tissue shear stiffness will be measured in the right hepatic lobe [in kilopascals (kPa)] to assess the degree of fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Walker, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Morningside, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  To achieve aims in the approved proposal. Proposals should be directed to ryan.walker@mssm.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years.